CLINICAL TRIAL: NCT02211625
Title: A Two-Part Study to Evaluate the Safety, Tolerability, Pharmacodynamics And Pharmacokinetics of TRV734 in Healthy Adult Male and Female Subjects
Brief Title: A Safety, Tolerability, PD and PK Study in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP734-1002
Record Dates: First submitted 2014-07-29; First posted 2014-08-07 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Healthy; Pharmacodynamics (PD); Pharmacokinetics (PK)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRV734 125 mg (Experimental): Part A, open-label will evaluate the the safety, PK and PD profile of a 125mg dose of TRV734 in which subjects are fasted, fed a standard meal, or fed a high-fat meal. Part A will also inform the dosing paradigm for Part B.
  Interventions: Drug: Open-label TRV734 125 mg
- Multiple ascending dose study, active and placebo comparators (Active Comparator): Part B will assess the safety, tolerability, PD and PK of TRV734. Subjects will be randomized in a ratio of 3:1:1 to receive either multiple doses of TRV734, oxycodone IR 10mg or placebo.
  Interventions: Drug: TRV734 blinded; Drug: Oxycodone IR 10 mg; Drug: Placebo

INTERVENTIONS:
Drug: Open-label TRV734 125 mg — 125 mg
  Arms: TRV734 125 mg
Drug: TRV734 blinded — blinded, multiple ascending dose
  Arms: Multiple ascending dose study, active and placebo comparators
Drug: Oxycodone IR 10 mg
  Arms: Multiple ascending dose study, active and placebo comparators
Drug: Placebo — TRV734-matched and oxycodone placebo
  Arms: Multiple ascending dose study, active and placebo comparators

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of TRV734 given as a single dose (Part A) and as multiple ascending doses (Part B) in healthy subjects.

DETAILED DESCRIPTION:
This will be conducted in two-parts enrolling a total of approximately 72 healthy volunteers.

* Part A will assess the safety, tolerability, PD and PK of a 125mg dose of TRV734 in an open-label, randomized, three-period crossover study in which subjects are fasted, fed a standard meal, or fed a high-fat meal.
* Part B of the trial will assess the safety, tolerability, PD and PK of multiple ascending doses of TRV734 in a double blind, double dummy, randomized, active- and placebo-controlled, adaptive study. Oxycodone immediate release (IR) 10 mg will be used as a benchmark.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician or trained qualified designee
* Males (Part A) or males and females (Part B) between 18 & 64 years of age, inclusive. Females must be of non-childbearing
* Capable of giving written informed consent

Exclusion Criteria:

* Clinically significant conditions, or history of fainting or syncope
* Medical or psychiatric illness
* Major surgery within 4 weeks of screening
* Known difficulty with obtaining intravenous access
* Any ophthalmologic condition that could interfere with pupillometry
* History of sensitivity to any of the investigational products, or known intolerance to opioids or a history of medication or other allergy
* Use of prescription or non prescription medications
* History of drug abuse within 6 months of screening
* Use of any illegal drug within 30 days of screening and throughout participation in the study
* History of smoking or use of nicotine containing products within 3 months of screening and throughout participation in the study
* Donation of blood or plasma within 4 weeks prior to dosing
* Participation in a clinical trial and has received a medication within 30 days
* Weight <50 kg or BMI outside range of 18 - 32 kg/m2
* Positive for HIV antibody, hepatitis B virus surface antigen, or hepatitis C virus
* If male, unwillingness to abstain from sexual intercourse with a pregnant or lactating woman and, if engaging in sexual intercourse with a female partner of childbearing potential, use a condom and spermicide, in addition to having their female partner use another form of contraception, and abstain from sperm donation
* Part B Only:

  * Active dermatological condition or eczema on non-dominant hand.
  * Peripheral vascular disease
  * If female, of child bearing potential, pregnant or breastfeeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety | 7 days
  Clinical safety data from adverse event reporting, clinical observations, 12-lead ECGs, cardiac telemetry monitoring, vital signs (blood pressure, heart rate, respiratory rate and oral temperature), oxygen saturation and safety laboratory tests.

SECONDARY OUTCOMES:
Effect on pharmacodynamics of multiple ascending doses (Part B) of TRV734 | 4 days
  Change from baseline in: Pupillometry and Cold Pain Test
Effect on pharmacokinetics of multiple ascending (Part B) doses of TRV734 | 4 days
  From the plasma concentration-time data, the following PK parameters will be determined, as data permit: AUC, Cmax, tmax, t½,eff, Vss/F, C, AR, and CL/F. From the urine concentration data, the following will PK parameters will be determined, as data permit: %UR and CLR.
Effect on pharmacodynamics of 125mg dose or TRV734 (Part A) following various administration paradigms | 7 days
  Change from baseline in: Pupillometry and Cold Pain Test
Effect on pharmacokinetics of 125mg dose of TRV734 (Part A) following various administration paradigms. | 7 days
  From the plasma concentration-time data, the following PK parameters will be determined, as data permit: AUC, Cmax, tmax, t½,eff, Vss/F, C, AR, and CL/F. From the urine concentration data, the following will PK parameters will be determined, as data permit: %UR and CLR.

CONTACTS AND LOCATIONS:
Overall Officials: Franck Skobieranda, MD, Study Director — Trevena Inc.
Locations (1):
- ICON Development Solutions, San Antonio, Texas, United States